CLINICAL TRIAL: NCT00613223
Title: Phase I Dose Escalation of Vandetanib (Zactima, ZD6474) in Combination With Etoposide for Malignant Gliomas
Brief Title: Ph I Dose Escalation Trial of Vandetanib in Combo w Etoposide for Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annick Desjardins (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assist Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001919
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Gliosarcoma; Glioblastoma
Keywords: Malignant Gliomas; Etopophos; Toposar; VePesid; Etoposide; Vandetanib; Zactima; ZD6474; VP-16; Brain Tumor; Recurring Malignant Brain Tumor; Gliosarcoma; Glioblastoma; Glioma; Malignant Glioma; GBM
MeSH Terms: conditions — Gliosarcoma; Glioblastoma; Glioma; Brain Neoplasms | interventions — vandetanib; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib and Etoposide (Experimental): Patients will be stratified based on whether they are receiving an enzyme-inducing anti-epileptic drug (EIAED). The dose level of vandetanib will be increased in successive cohorts of subjects. Etoposide will be given daily at a dose of 50 mg/ day for 21 days followed by 7 days with no etoposide.
  Interventions: Drug: Vandetanib and Etoposide

INTERVENTIONS:
Drug: Vandetanib and Etoposide — Vandetanib will be given orally once day. Swallow tablet with 240 ml of non-carbonated water. Initial dose is 100 mg/day for stratum 1 & 200 mg/day for stratum 2. Etoposide will be taken by mouth in capsule form at a flat dose of 50 mg/day for 1st 21 days of 28-day cycle. You will not take etoposide for following 7 days of the cycle.
  Other Names: Vandetanib - Zactima (ZD 6474); Etoposide - VP-16, Etopophos, Toposar, VePesid

SUMMARY:
Primary Objective: To determine maximum tolerated dose & dose limiting toxicity of vandetanib when combined with standard dosing of etoposide among patients with recurrent malignant glioma who are on & not on enzyme-inducing anti-epileptic drugs (EIAEDs) Secondary Objectives: To assess safety & tolerability of vandetanib + etoposide in this population; To evaluate pharmacokinetics of vandetanib among malignant glioma patients on & not on EIAEDs when combined with etoposide.

Exploratory Objective: To evaluate for evidence of anti-tumor activity of study regimen among recurrent malignant glioma patients including radiographic response rate, 6-month progression free survival (PFS) rate & median PFS.

DETAILED DESCRIPTION:
This is open-label, single center, 2-cohort phase I dose-escalation study of vandetanib administered orally on continuous daily dosing schedule + oral etoposide among adult patients with recurrent or relapsing malignant glioma. Patients will be stratified based on whether they are receiving EIAEDs & each stratum will independently dose escalate. Dose of vandetanib will be increased in successive cohorts of patients. Etoposide will be given daily at a dose of 50mg/day for 21 days followed by 7 days with no etoposide. Cohorts of 3-6 subjects will accrue at each dose level until maximum tolerated dose (MTD) is defined. Subjects will be adult patients with histologically confirmed malignant glioma who are presenting at time of recurrence/relapse. Up to 48 subjects will be enrolled.

Sample size will be based on modified, classical "3+3" dose escalation design. Primary safety & efficacy analysis will be conducted on all subject data at time all subjects who are still receiving study drug will have completed at least 4 cycles of treatment. Most common adverse events (AEs) associated with vandetanib are rash, diarrhea, & asymptomatic QTc prolongation. Protracted oral dosing of etoposide is associated with toxicity that is mild in most patients & consists mainly of myelosuppression & diarrhea. Less commonly, protracted etoposide dosing has been associated w more significant hematologic toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients have baseline evaluations ≤14days prior to 1st dose of study drug unless otherwise specified

* Patients with confirmed malignant glioma (MG) who are recurrence/relapse
* Patients may not have stereotactic tumor biopsy < 1 week or surgical resection or open biopsy < 4 weeks before starting study drug
* For stratum of non-EIAED patients, each patient must be off all EIAEDs for > 2 weeks prior to starting study drug; similarly for stratum of EIAED patients, each patient must be on EIAED for >2 weeks prior to starting study drug
* Patients should be on non-increasing dose of steroids for >7 days prior to obtaining baseline MRI with gadolinium (Gd-MRI) of brain
* Patients should be on non-increasing dose of steroids for >7 days prior to starting study drug
* Multifocal disease is eligible
* Age ≥ 18 years
* Karnofsky Performance Status (KPS) ≥70
* Absolute Neutrophil Count ≥1.0 x 10 9/L
* Hemoglobin (Hgb) ≥9 g/dL
* Platelets ≥100 x 10 9/L
* Serum creatinine ≤1.5 x ULRR or measured 24-hr CrCl ≥50mL/min/1.73m2
* Life expectancy ≥ 12 weeks
* Written informed consent obtained prior to screening procedures
* Negative Beta-HCG pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Laboratory Results:
* Serum direct bilirubin >1.5 x upper limit of normal (ULN) of reference range
* Serum creatinine >1.5 x ULRR & CrCl <30 mL/min
* Potassium, <4.0 mmol/L despite supplementation; serum calcium, magnesium out of normal range despite supplementation
* ALT or AST > 2.5 x ULRR
* Evidence of severe/uncontrolled systemic disease or any concurrent condition which in Investigator's opinion makes it undesirable for patient to participate in trial or which would jeopardize compliance with protocol
* Clinically significant cardiovascular event such as myocardial infarction, superior vena cava syndrome, New York Heart Association classification of heart disease >2 within 3 months before entry; or presence of cardiac disease that, in opinion of Investigator, increases risk of ventricular arrhythmia
* History of arrhythmia which is symptomatic/requires treatment/asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
* Previous history of QTc prolongation as result from other medication that required discontinuation of that medication
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death <40 years
* Presence of left bundle branch block
* QTc with Bazett's correction that's unmeasureable, or ≥ 480msec on screening EEG.
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes/induce CYP3A4 function except for EIAEDs
* Hypertension not controlled by medical therapy
* Currently active diarrhea that may affect ability of patient to absorb study regimen/tolerate diarrhea
* Women who are currently pregnant/breast feeding
* Previous or current malignancies of other histologies the last year, with exception of cervical carcinoma in situ & adequately treated basal cell or squamous cell carcinoma of skin
* Receipt of any investigational agents <30 days prior to commencing study treatment unless pt has recovered from all anticipated toxicities of investigational agent
* Last dose of prior chemo discontinued < 4 weeks before start of study therapy unless pt has recovered from all anticipated toxicities of chemo
* Last XRT < 4 weeks before start of study therapy, unless patient has recovered from all anticipated toxicities of XRT
* Any unresolved toxicity >CTC gr1 from previous anti-cancer therapy
* Previous enrollment/randomization of treatment in present study
* Major surgery < 4 weeks/incompletely healed surgical incision before starting study therapy
* Patients who have received prior oral VEGFR, EGFR or PDGFR-directed therapies. Patients who received prior Avastin will be eligible as long as at least 6 weeks has elapsed since last dose.
* Patients taking warfarin sodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, biologic activity, & pharmacokinetic profile of vandetanib when used in combo w etoposide | 6-month progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/